CLINICAL TRIAL: NCT06015971
Title: Omega-3 Enriched Supplements in the Nutritional Support of Patients With Gastrointestinal Cancer
Brief Title: Omega-3 Fatty Acids and Nutritional Support in Gastrointestinal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Sarcopenia omega3
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia
Keywords: cancer; nutritional support; omega-3 enriched nutritional supplements
MeSH Terms: conditions — Sarcopenia; Neoplasms | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard hypercaloric, hyperproteic oral supplement (Active Comparator)
  Interventions: Dietary Supplement: Standard
- omega-3 enriched oral supplement (Experimental)
  Interventions: Dietary Supplement: omega-3

INTERVENTIONS:
Dietary Supplement: omega-3 — Take 2 omega-3 enriched oral supplements per day plus physical activity and Mediterranean Diet
  Arms: omega-3 enriched oral supplement
Dietary Supplement: Standard — Take 2 hypercaloric hyperproteic oral supplements per day plus physical activity and Mediterranean Diet
  Arms: standard hypercaloric, hyperproteic oral supplement

SUMMARY:
Sarcopenia is a frequent complication in patients with cancer and chronic diseases, it is characterized by decreased muscle strength and fatigue due to reduced skeletal muscle mass, which is accompanied by atrophy and decreased quality of muscle tissue. In all cases, it negatively impacts treatment tolerance, clinical outcomes and survival, in consequence, quality of life of these patients decreases while morbidity, mortality and costs increase. In this context, appropriate nutritional screening and early nutrition support are extremely recommended, to this aim, in some cases, oral nutritional supplements (ONS) are necessary; ONS could have a standard formula or be enriched with specific nutrients (arginine, glutamine, branched chain amino acids, n-3 fatty acids, and nucleotides), which can modulate the activity of the immune system and provide an additional benefit beyond the nutritional support, this intervention type is called immunonutrition. Despite these possible benefits, their utility has been proven in few clinical scenarios, for example in with patients with upper gastrointestinal cancer undergoing surgical resection; based on this, current guidelines recommend that patients should receive oral/enteral nutritional support with an specific formula enriched in immunonutrients (with arginine, n-3 fatty acids or nucleotides) , but there is a lack of evidence for supporting its use in other clinical conditions including patients with cancer that receive systemic treatment

ELIGIBILITY:
Inclusion Criteria:

* - Patients with Gastrointestinal tumor undergoing systemic treatment (chemo-radio-immuno therapy or their combination)
* Body weight loss >5% in the previous three months or >10% in the previous six months
* Both sexes
* Age between 18-85 y-old.

Exclusion Criteria:

* Life expectancy < 2 weeks
* MDRD < 15 mL/min
* End-stage liver disease
* Any musculoskeletal, cardiovascular and/or neurological disorders that could affect exercising.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | 12 weeks
  Muscle mass change (in Kg)
Functionality | 12 weeks
  Changes in functionality measured with the Up and Go Test

SECONDARY OUTCOMES:
Albumin | 12 weeks
  Changes in serum albumin levels (g/dl)
C-RP | 12 weeks
  Changes in serum C-RP(g/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- IMIBIC, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided